CLINICAL TRIAL: NCT02982031
Title: A Comparison of Visualization Between Shamrock Technique and Paramedian Transverse Scan in Lumbar Plexus Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 302/2559(EC4)
Record Dates: First submitted 2016-09-18; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Lumbar Plexus Blockade
Keywords: Ultrasound-guided lumbar plexus blockade; Shamrock technique; Paramedian transverse scan; USG LPB; USGRA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- shamrock (Sham Comparator): shamrock: both left and right sided scan,both intertransverse and transverse process window
  Interventions: Procedure: shamrock
- paramedian transverse scan (Active Comparator): paramedian transverse scan (PMTS): both left and right, both intertransverse and transverse process window
  Interventions: Procedure: paramedian transverse scan

INTERVENTIONS:
Procedure: shamrock — This scanning technique is performed in the lateral decubitus position with the side of interest facing upwards. The transducer is placed in the transverse plane on the flank of the patient cranially to the iliac crest. The quadratus lumborum muscle is identified medial to the aponeurosis of the transversus abdominis muscle. With the psoas muscle anterior to the transverse process, the erector spinae muscle posterior to the transverse process, and the quadratus lumborum muscle attached to the apex of the transverse process of L4.
  Arms: shamrock
Procedure: paramedian transverse scan — The ultrasound transducer is positioned 4 cm lateral to the midline along the intercristal line and just above the iliac crest. The transducer is also directed slightly medially.
  Arms: paramedian transverse scan

SUMMARY:
The primary objective of this study was to compare ultrasound visibility of the lumbar plexus at the intertransverse space between paramedian transverse scan and shamrock technique. Moreover obtaining a clear image of relevant structures is imperative. Thus, the secondary objective was to assess ultrasound visibility of each relevant structure and overall visibility between these two methods.

DETAILED DESCRIPTION:
Background: Ultrasound-guided lumbar plexus block (USG LPB) is regarded as a form of advanced ultrasound-guided regional anesthesia (USGRA). One of the key challenges of USG LPB is visualization of the lumbar plexus. That are currently in use for ultrasound-guided lumbar plexus blockade - paramedian transverse scan (PMTS) and shamrock technique.

Method: Twenty-three healthy adult volunteers aged ≥ 18 years were enrolled in this prospective cohort study. Ultrasound visualization results were compared between methods.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer, age >/= 18

Exclusion Criteria:

* spinal deformity and history of previous back or spine surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Video (VDO) loops visualization of lumbar plexus | 1 month
  Percentage of Video (VDO) loops visualization of lumbar plexus comparing between two techniques

SECONDARY OUTCOMES:
Ultrasound visibility score of each relevant structures | 1 month
  10 structures: Erector spinae muscle, Quadratus lumborum muscle, Psoas muscle, Vertebral body, Inferior vena cava, Articular process of the lumbar vertebra, Lumbar paravertebral space, lumbar nerve root, Lumbar plexus nerve, Psoas compartment Using 4-point Likert scale (0, not visible; 1, hardly visible; 2, well visible; 3, very well visible)
Overall ultrasound visibility score of 10 structures | 1 month
  Sum of ultrasound visibility score of 10 relevant structures: Erector spinae muscle, Quadratus lumborum muscle, Psoas muscle, Vertebral body, Inferior vena cava, Articular process of the lumbar vertebra, Lumbar paravertebral space, lumbar nerve root, Lumbar plexus nerve, Psoas compartment

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pawinee, M.D, Principal Investigator — 66864001721
Locations (1):
- Siriraj hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No